CLINICAL TRIAL: NCT03986450
Title: The Impact of Implementing ERAS Protocol on Healthcare Costs in Patients Undergoing Laparoscopic Hysterectomy
Brief Title: ERAS Protocol in Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aysu Akca, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AYSUAKCA2
Record Dates: First submitted 2019-05-23; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Surgery
Keywords: Enhanced recovery after surgery; Laparoscopic hysterectomy
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Active Comparator): Patients in this group will receive ERAS protocol preoperatively, perioperatively and postoperatively.
  Interventions: Other: Enhanced recovery after surge(ERAS) protocol
- Control (No Intervention): This group of patients will not receive ERAS care and will undergo a standard laparoscopic hysterectomy.

INTERVENTIONS:
Other: Enhanced recovery after surge(ERAS) protocol — The components of ERAS multidisciplinary pathway concerning preoperative, operative, and postoperative period are as follows:
  1. Preoperative care:
     Counseling before hospital admission Fluid, and carbohydrate loading Avoiding prolongation of the fasting period Avoiding bowel preparation or its application only in selective cases Application of antibiotic prophylaxis Application of thromboprophylaxis
  2. Perioperative care:
  Use of short-acting anesthetic agents Application of midthoracic, epidural anesthesia/analgesia Refraining from using drains Refraining from salt, and water overload Maintenance of normothermia
  Postoperative care:
  Application of midthoracic, epidural anesthesia/analgesia Prevention of nausea, and vomiting Refraining from salt, and water overload Earlier removal of catheters Initiation of oral intake at an early period Use of nonopioid oral analgesics/NSAIDs Early mobilization
  Arms: ERAS group

SUMMARY:
ERAS protocol has been shown to improve patient comfort and reduce the length of hospital stay. This study aimed to investigate the impact of implementing ERAS protocols on healthcare costs in patients undergoing a laparoscopic hysterectomy.

DETAILED DESCRIPTION:
ERAS protocol has been shown to improve patient comfort and reduce the length of hospital stay in various kinds of surgical procedures. This study aimed to investigate whether ERAS protocol has an impact on healthcare costs in patients undergoing a laparoscopic hysterectomy. Patients scheduled for laparoscopic hysterectomy will be allocated to one of the study groups: ERAS group patients will receive ERAS protocol during the perioperative period; Conventional care groups will undergo standard abdominal hysterectomy without the implementation of ERAS protocol. The groups will be compared with respect to the length of hospital stay, rehospitalizations, and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for laparoscopic hysterectomy

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) class IV
* Development of complications during surgery
* Body mass index > 40 kg/m2

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-07-18 (Estimated)

PRIMARY OUTCOMES:
Healthcare costs | Up to one month
  Hospital costs will be obtained from the accounting office of the hospital

SECONDARY OUTCOMES:
Length of stay | Up to one month
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Aysu Akca, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Department of Obstetrics and Gynecology, University of Health Sciences, Faculty of Medicine, Kanuni Sultan Suleyman Hospital,, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No